CLINICAL TRIAL: NCT06185231
Title: Investigation of the Effects of Percussion Massage Therapy After Anterior Cruciate Ligament Injury
Brief Title: Investigation of the Effects of Vibration Therapy on Pain, Functionality, and Proprioception After ACL Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, burak menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-772.02-6782
Record Dates: First submitted 2023-11-28; First posted 2023-12-29 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Vibration Therapy; Anterior Cruciate Ligament Injuries
Keywords: Vibration; Anterior Cruciate Ligament; joint position sense
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percussion Massage Group (Experimental): Both groups will undergo a progressive exercise program given as Phase-1, Phase-2, and Phase-3 for 6 weeks. The Percussion massage group will receive percussion massage therapy for a total of 5 minutes for each muscle group.The application will be done to the Quadriceps and Hamstring muscle groups before exercise. The device will be used with a soft connection head at 33-40 Hz. A total of 5 minutes of percussion massage will be applied to each muscle group. In the first 2.5 minutes of the massage therapy, the medial side of the focus muscle will be targeted, and in the second 2.5 minutes, the lateral side of the focus muscle will be targeted. Neuromuscular Electrical Stimulation (NMES) will be applied to the Quadriceps muscle group for facilitation and reeducation purposes.
  Interventions: Other: Percussion Massage Group
- Conventional Group (Active Comparator): Conventional group undergo a progressive exercise program given as Phase-1, Phase-2, and Phase-3 for 6 weeks.
  Neuromuscular Electrical Stimulation (NMES) will be applied to the Quadriceps muscle group for facilitation and reeducation purposes.
  NMES Parameters:
  Electrode placement: will be applied to motor points and the muscle belly to achieve optimal contraction.
  Frequency: 50-70 Hz Duration: 20 minutes.
  Interventions: Other: Conventional Group

INTERVENTIONS:
Other: Percussion Massage Group — In addition progressive exercise program, The Percussion massage group will receive percussion massage therapy for a total of 5 minutes for each muscle group. The application will be done to the Quadriceps and Hamstring muscle groups before exercise. Neuromuscular Electrical Stimulation (NMES) will be applied to the Quadriceps muscle group for facilitation and reeducation purposes.
  Arms: Percussion Massage Group
Other: Conventional Group — Conventional group undergo a progressive exercise program given as Phase-1, Phase-2, and Phase-3 for 6 weeks.
  Neuromuscular Electrical Stimulation (NMES) will be applied to the Quadriceps muscle group for facilitation and reeducation purposes.
  Arms: Conventional Group

SUMMARY:
Over the past decade, vibration therapy has gained popularity. This treatment involves the transmission of vibration either through whole-body vibration (WBV) platforms or by applying local vibration (LV) directly to the muscles or tendons. In the context of ACLR (anterior cruciate ligament reconstruction), it has been reported that a single session of either WBV or LV, applied while patients maintain a squatting position, acutely improves the strength of the Quadriceps muscle when applied 50 months post-surgery, possibly by reducing arthrogenic muscle inhibition. Another study tested whether local vibration training (LVT) in the early post-ACLR phase (first 10 weeks) could improve strength recovery and found that LVT enhances strength regain after ACLR. This feasibility study demonstrates that LVT applied to relaxed muscles is a promising method of vibration therapy that can be applied early in ACLR. Compared to traditional massage, vibration therapy may also improve strength parameters.

Percussion massage therapy is a new method that combines elements of traditional massage and vibration therapy. In the literature, there is a lack of scientific evidence on how and to what extent percussion massage therapy affects range of motion (ROM) and muscle strength. To date, only one conference paper has investigated the effects of a handheld percussion massage therapy device, and they found no change in vertical jump height after a 5-minute percussion massage therapy session applied to several lower body muscle groups." A review of the literature reveals that to date, there has been no study investigating the effects of manually applied percussion massage therapy on pain, functionality, and proprioception in cases who have undergone anterior cruciate ligament surgery. Therefore, the purpose of our study is to examine the effects of percussion massage therapy on pain, joint range of motion, joint position sense, muscle diameter, balance parameters, and functionality in patients who have undergone surgery following an anterior cruciate ligament injury.

DETAILED DESCRIPTION:
The study will be conducted at Medipol University Hospital.The study will include 30 individuals aged 20-40 who have undergone anterior cruciate ligament surgery and subsequently presented to the physical therapy outpatient clinic. All participants will be informed about the study and asked to sign a voluntary consent form. Assessments will be applied to all participants. Inclusion Criteria: Having a hamstring tendon autograft, allograft, or undergone anterior cruciate ligament reconstruction Complete unilateral ACL rupture Applying to the physical therapy clinic within the first two weeks after surgical reconstruction Being in the age range of 20-40 Agreeing to participate in the study Having signed the informed consent form Exclusion Criteria: Presence of other intra-articular and extra-articular ligament/cartilage pathology in addition to the ACL rupture History of secondary reconstruction surgery Diagnosis of specific mechanical (alignment) disorder of the lower extremity Presence of central and peripheral nervous system diseases Diseases affecting the musculoskeletal, neurological, and vestibular systems Presence of chronic and systemic diseases that may cause peripheral neuropathy and loss of deep sensation (e.g., diabetes, chronic kidney failure) Presence of cognitive, mental, and psychological problems Presence of balance problems or use of medication that negatively affects balance History of accompanying autoimmune or inflammatory diseases such as rheumatoid arthritis, lupus erythematosus." Participants will consist of individuals referred by Physical Medicine and Rehabilitation physicians at Medipol University Esenler Hospital to a physiotherapist to receive physical therapy after anterior cruciate ligament surgery. The demographic information of the participants (name, age, gender, marital status, education level, profession, dominant side, affected side, duration of pain, history of surgical operation) will first be inquired. Then, pain, joint range of motion, joint position sense, muscle diameter measurement, and balance parameters will be evaluated.

The evaluation methods will be applied to the participants before and after the treatment.

In patients who have undergone anterior cruciate ligament surgery;

* Proprioception > Joint Position Sense (Goniometer Pro)
* Pain > Visual Analog Scale
* Balance > Berg Balance Scale
* Functionality > Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
* Joint Range of Motion > Goniometer Pro
* Quality of Life > Short Form-36 will be measured.

Smartphone Application Goniometer Pro For knee joint range of motion assessment with a smartphone, subjects are positioned prone. The smartphone is placed on the lateral midline of the tibia to establish 0° knee joint extension, then active knee flexion is performed, and angular data is obtained, followed by passive knee flexion performed by the practitioner and angular data is taken again.

Assessment of Joint Position Sense For the assessment of knee joint position sense, the starting position is considered as 90° flexion. For the first target angle of 60° knee flexion, the physiotherapist passively brings the patient's knee to 60° knee flexion, holds it in that position for 5 seconds, and asks the patient to remember this angle and say "here" when they think they have reached this angle during the test. The physiotherapist returns the patient's knee to the starting position of 90° knee flexion and asks the patient to rest in the starting position for 5 seconds. Before proceeding with the test, the target angle is repeated 3 times with eyes open and 3 times with eyes closed, and the patient's "perceived target angle" in degrees is recorded. The test for one target angle is repeated 6 times by the patient and the average of 6 measurements is recorded. In the assessment of joint position sense, the patient's estimated angle is considered the actual value, and the deviation from the target angle is considered as the absolute error.

Visual Analog Scale (VAS) The Visual Analog Scale is used to measure the intensity of pain. The patient is asked to assess their pain on a line with values ranging from 0-10, where 0 means no pain, and 10 means unbearable pain. Individuals mark their pain intensity on this line according to their pain situation.

Berg Balance Scale The scale includes 14 different activities assessing functions such as getting up from sitting, sitting without support, standing without support, sitting while standing, standing with eyes closed, transfers, standing with legs together, picking up objects from the floor, reaching forward while standing, looking back while turning, turning 360 degrees, standing on a stable side stool, standing with one foot in front, and standing on one foot. Each activity is scored between 0-4. The scoring of the scale is done by adding up the scores from each section. According to the results obtained from the scale; ≤20 indicates wheelchair level, >20≤40 indicates walking with assistance, and >40≤56 indicates independence.

Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) The scale is a valid and reliable measure used to assess physical function in patients who have undergone knee surgery. The scale consists of a total of 24 questions: 5 questions related to pain (0-20 points), 2 questions related to stiffness (0-8 points), and 17 questions related to physical function difficulty (0-68 points). Higher WOMAC scores indicate a greater degree of impairment.

Short Form-36 (SF-36) It is a 36-item questionnaire containing eight domains measuring physical and mental components (PCS and MCS, respectively). Each item is scored and totaled according to a standard scoring protocol. Each domain is scored between 0 to 100. Higher scores indicate a better health status."

ELIGIBILITY:
Inclusion Criteria:

* Having a hamstring tendon autograft, allograft, or undergone anterior cruciate ligament reconstruction Complete unilateral ACL rupture
* Applying to the physical therapy clinic within the first two weeks after surgical reconstruction
* Being in the age range of 20-40
* Agreeing to participate in the study
* Having signed the informed consent form

Exclusion Criteria:

* Presence of other intra-articular and extra-articular ligament/cartilage pathology in addition to the ACL rupture
* History of secondary reconstruction surgery
* Diagnosis of specific mechanical (alignment) disorder of the lower extremity
* Presence of central and peripheral nervous system diseases
* Diseases affecting the musculoskeletal, neurological, and vestibular systems
* Presence of chronic and systemic diseases that may cause peripheral neuropathy and loss of deep sensation (e.g., diabetes, chronic kidney failure)
* Presence of cognitive, mental, and psychological problems
* Presence of balance problems or use of medication that negatively affects balance
* History of accompanying autoimmune or inflammatory diseases such as rheumatoid arthritis, lupus erythematosus.

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Range of motion | Baseline
  For knee joint range of motion assessment with a smartphone, subjects are positioned prone. The smartphone is placed on the lateral midline of the tibia to establish 0° knee joint extension, then active knee flexion is performed, and angular data is obtained, followed by passive knee flexion performed by the practitioner and angular data is taken again.
Joint Position Sense | Baseline
  For the assessment of knee joint position sense, the starting position is considered as 90° flexion. For the first target angle of 60° knee flexion, the physiotherapist passively brings the patient's knee to 60° knee flexion, holds it in that position for 5 seconds, and asks the patient to remember this angle and say "here" when they think they have reached this angle during the test. The physiotherapist returns the patient's knee to the starting position of 90° knee flexion and asks the patient to rest in the starting position for 5 seconds. Before proceeding with the test, the target angle is repeated 3 times with eyes open and 3 times with eyes closed, and the patient's "perceived target angle" in degrees is recorded.
Visual Analog Scale | Baseline
  The Visual Analog Scale is used to measure the intensity of pain. The patient is asked to assess their pain on a line with values ranging from 0-10, where 0 means no pain, and 10 means unbearable pain. Individuals mark their pain intensity on this line according to their pain situation.
Berg Balance Scale | Baseline
  The scale includes 14 different activities assessing functions such as getting up from sitting, sitting without support, standing without support, sitting while standing, standing with eyes closed, transfers, standing with legs together, picking up objects from the floor, reaching forward while standing, looking back while turning, turning 360 degrees, standing on a stable side stool, standing with one foot in front, and standing on one foot. Each activity is scored between 0-4. The scoring of the scale is done by adding up the scores from each section. According to the results obtained from the scale; ≤20 indicates wheelchair level, >20≤40 indicates walking with assistance, and >40≤56 indicates independence.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index | Baseline
  The scale is a valid and reliable measure used to assess physical function in patients who have undergone knee surgery. The scale consists of a total of 24 questions: 5 questions related to pain (0-20 points), 2 questions related to stiffness (0-8 points), and 17 questions related to physical function difficulty (0-68 points). Higher WOMAC scores indicate a greater degree of impairment.
Short Form-36 | Baseline
  It is a 36-item questionnaire containing eight domains measuring physical and mental components (PCS and MCS, respectively). Each item is scored and totaled according to a standard scoring protocol. Each domain is scored between 0 to 100. Higher scores indicate a better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Menek, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Erayata BN, Menek B. Investigating the effects of percussion massage therapy on pain, functionality, muscle diameter, and proprioception in individuals with ACL reconstruction: a randomized controlled trial. PLoS One. 2025 Mar 26;20(3):e0319731. doi: 10.1371/journal.pone.0319731. eCollection 2025. PMID 40138389